CLINICAL TRIAL: NCT01649817
Title: Multicenter REtrospective Study to Evaluate coMpliance to Therapy and Drug survIval of Tocilizumab (TCZ) in patientS With Moderate to Severe actIve rheumatOid Arthritis in routiNe Daily Clinical Practice (REMISSION II Study)
Brief Title: A Retrospective Observational Study on Compliance in Patients With Rheumatoid Arthritis on Treatment With RoActemra/Actemra (Tocilizumab) in Clinical Practice (REMISSION II)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28258
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, retrospective observational study will evaluate compliance an reasons for withdrawal in patients with moderate to severe active rheumatoid arthritis on treatment with intravenous RoActemra/Actemra (tocilizumab) in daily clinical practice. Data will be collected from each eligible patient over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised 1987 ACR criteria at baseline
* RoActemra/Actemra treatment must have been initiated 6 months prior to ICF signing
* Patient eligible according to the summary of product characteristics (SPC) and routine clinical practice/European recommendations for the use of biologic DMARDs for the treatment of rheumatoid arthritis

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* Participation in interventional clinical trials during the observational period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients suitable for treatment with RoActemra/Actemra according to SPC
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients on RoActemra/Actemra at 6 months after initiating treatment | 12 months

SECONDARY OUTCOMES:
Frequency of withdrawal (according to reasons) | 12 months
Frequency of dose modifications | 12 months
Change in disease activity (DAS28) | from baseline to Month 6 or withdrawal, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Greece (17):
  - Agios Dimitrios
  - Agía Paraskeví
  - Argiroupoli
  - Athens
  - Chalandri
  - Chania
  - Corinth
  - Eleusina
  - Herakleio
  - Ioannina
  - Kifissia
  - Peristeri
  - Peuki
  - Rethymno
  - Serres
  - Thessaloniki
  - Volos